CLINICAL TRIAL: NCT00004646
Title: Phase III Randomized, Double-Blind Study of Prednisone for Duchenne Muscular Dystrophy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); University of Rochester (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: 199/11695; URMC-2251
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-12

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Duchenne muscular dystrophy; genetic diseases and dysmorphic syndromes; muscular dystrophy; neurologic and psychiatric disorders; rare disease
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Genetic Diseases, Inborn; Muscular Dystrophies; Neurologic Manifestations; Mental Disorders; Rare Diseases | interventions — Prednisone

INTERVENTIONS:
Drug: prednisone

SUMMARY:
OBJECTIVES: I. Characterize the effect of prednisone on muscle protein metabolism in patients with Duchenne muscular dystrophy.

II. Determine whether prednisone changes levels of insulin-like growth factor 1, growth hormone, and insulin.

III. Characterize the effect of prednisone on muscle morphometry and muscle localization of utrophin.

IV. Compare the prednisone response in patients with Duchenne muscular dystrophy to that seen in normal individuals and in patients with facioscapulohumeral dystrophy.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, double-blind study. Patients are randomly assigned to prednisone or placebo. Therapy is administered daily for 12 weeks; prednisone is then tapered.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

* Ambulatory males with Duchenne muscular dystrophy
* No medical/psychiatric contraindication to protocol therapy
* No requirement for regular use of prescription medication

Ages: 5 Years to 15 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20
Dates: Start 1995-04

CONTACTS AND LOCATIONS:
Overall Officials: Robert Griggs, Study Chair — University of Rochester